CLINICAL TRIAL: NCT01808287
Title: Safety and Performance Study of the Edwards SAPIEN 3 Transcatheter Heart Valve
Brief Title: Safety and Performance Study of the Edwards SAPIEN 3 Transcatheter Heart Valve/ The SAPIEN 3 Study
Acronym: SAPIEN3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-07
Record Dates: First submitted 2013-03-07; First posted 2013-03-11 (Estimated); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Aortic Valve Disease
Keywords: Transcatheter Aortic Valve Replacement; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High risk population (Experimental): SAPIEN 3 transcatheter heart valve was implanted in high risk patients
  Interventions: Device: Edwards SAPIEN 3 Transcatheter Heart Valve
- Intermediate risk population (Experimental): SAPIEN 3 transcatheter heart valve was implanted in intermediate risk patients
  Interventions: Device: Edwards SAPIEN 3 Transcatheter Heart Valve

INTERVENTIONS:
Device: Edwards SAPIEN 3 Transcatheter Heart Valve — The Edwards SAPIEN 3 Transcatheter Heart Valve (THV) System is indicated for use in symptomatic patients (intermediate or higher operable risk) with severe aortic stenosis requiring aortic valve replacement (AVR).
  Other Names: TAVR; TAVI

SUMMARY:
The purpose of this study is to assess the safety and device success of the Edwards SAPIEN 3 Transcatheter Heart Valve (S3 THV) and the Edwards Commander and Certitude Delivery Systems in patients with symptomatic, severe aortic stenosis who are indicated for aortic valve replacement.

DETAILED DESCRIPTION:
This is a non-randomized, prospective, multicenter safety and device success study. Two hundred fifty (250) patients are planned to be enrolled at up to 20 participating investigational centers in Europe and Canada. Patient participation will last for a minimum of 5 years. Patients will be assessed at the following intervals: baseline, hospital discharge, 30 days, 1 year and annually thereafter for a minimum of 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Severe symptomatic calcific aortic valve stenosis with:

   1. High surgical risk: STS Score ≥ 8 or EuroSCORE ≥ 15 (first 50 patients),
   2. High to Intermediate surgical risk: STS Score ≥ 4 or EuroSCORE ≥ 10 (patients 51 to 150).
   3. Intermediate surgical risk: STS Score 4 to 8 or Logistic EuroSCORE 10 to 15 (subsequent patients); except for 20mm valve implants (STS Score > 4 or EuroSCORE ≥ 10).
2. Age ≥ 75 years
3. NYHA ≥ II
4. Heart team (including examining cardiac surgeon) agrees on eligibility including assessment that TAVR is appropriate.
5. Study patient has provided written informed consent to comply with all of the study procedures and follow-up visits.

Exclusion Criteria:

1. Non-calcified aortic valve
2. Acute myocardial infarction ≤ 30 days before the intended treatment
3. Untreated clinically significant coronary artery disease requiring revascularization.
4. Aortic valve is a congenital unicuspid or congenital bicuspid valve.
5. Mixed aortic valve disease (with predominant aortic regurgitation)
6. Preexisting bioprosthetic valve or ring in any position
7. For Intermediate Risk patients enrolled under inclusion criterion 1.c) patients with untreated pre-existing conduction disturbances (AV Block and Bundle Branch Block).

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 250 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
All-cause mortality rate | 30 days post-index procedure
  NAP

SECONDARY OUTCOMES:
safety endpoints(VARC II) | Discharge or 72 hours (whichever is longer), 30 days, 1 and 5 years post-index procedure.
  safety endpoints
  composite of mortality, and major complications including THV-related dysfunction major bleeds MI new conduction abnormality new onset of AF time-related valve safety composite of valve structural deterioration

CONTACTS AND LOCATIONS:
Overall Officials: John Webb, MD, Principal Investigator — St. Paul's Hospital Vancouver (Canada)
Locations (17):
- Canada (2):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Laval, Institut universitaire de cardiologie et de pneumologie de Quebec, Laval, Quebec
- France (4):
  - Massy, Institut Jacques Cartier, Massy
  - Paris, Hopital Bichat, Paris
  - CHU Charles Nicolle, Rouen
  - CHU Rangueil, Toulouse
- Germany (5):
  - Kerckhoff Heartcenter, Bad Nauheim
  - Universitatsklinik Koln, Cologne
  - Universitatsklinik Essen, Essen
  - Universitares Herzzentrum Hamburg GmbH, Hamburg
  - Stadtisches Klinikum Kalsruhe, Karlsruhe
- Policlinico Universitario, Padua, Italy
- United Kingdom (5):
  - Royal Victoria Hospital, Belfast
  - London St. Thomas's Hospital, London
  - King's College Hospital, London
  - Barts Health NHS Trust Hospital, London
  - Derriford Hospital, Plymouth

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Vahanian A, Urena M, Walther T, Treede H, Wendler O, Lefevre T, Spence MS, Redwood S, Kahlert P, Rodes-Cabau J, Leipsic J, Webb J. Thirty-day outcomes in patients at intermediate risk for surgery from the SAPIEN 3 European approval trial. EuroIntervention. 2016 Jun 12;12(2):e235-43. doi: 10.4244/EIJV12I2A37. PMID 27290682
- [Derived] Webb J, Gerosa G, Lefevre T, Leipsic J, Spence M, Thomas M, Thielmann M, Treede H, Wendler O, Walther T. Multicenter evaluation of a next-generation balloon-expandable transcatheter aortic valve. J Am Coll Cardiol. 2014 Dec 2;64(21):2235-43. doi: 10.1016/j.jacc.2014.09.026. Epub 2014 Nov 24. PMID 25456759